CLINICAL TRIAL: NCT05719909
Title: Cognitive Training to Enhance Depression Relief: Testing an Adjunct to Clinical Esketamine Treatment
Brief Title: Testing the Effectiveness of Cognitive Training Among Depressed Patients Receiving Esketamine Treatment
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Current unavailability of resources
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Rebecca Price, Associate Professor of Psychiatry and Psychology, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY22090145
Record Dates: First submitted 2023-01-20; First posted 2023-02-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive Training (Experimental): 8 sessions of web-based cognitive training
  Interventions: Behavioral: Cognitive Training
- Sham Training (Sham Comparator): 8 sessions of web-based sham training
  Interventions: Behavioral: Sham Training

INTERVENTIONS:
Behavioral: Cognitive Training — 8 sessions of web-based cognitive training
  Arms: Cognitive Training
Behavioral: Sham Training — 8 sessions of web-based sham training
  Arms: Sham Training

SUMMARY:
In a sample of patients already receiving esketamine treatment as part of their clinical care, this project seeks to test whether we can improve depression by introducing helpful information delivered by a computer-based training protocol. This work could ultimately lead to the ability to treat depression more efficiently and with broader dissemination by rapidly priming the brain for helpful forms of learning.

ELIGIBILITY:
Inclusion Criteria:

Any patient aged 18-80 in the esketamine clinic in the Center for Interventional Psychiatry. The clinic's extensive screening and eligibility criteria for esketamine treatment will not be altered in any way, other than imposing the study-specific age range and the two exclusion criteria below.

Exclusion Criteria:

1. Patients who do not expect to remain located in the Pittsburgh area for a minimum of 1 month beyond study enrollment.
2. Patients who, in the judgment of the esketamine clinical medical director, show signs of intellectual disability, developmental disability, and/or cognitive impairment (including age-related cognitive decline) of a sufficient degree to interfere with engagement in any study procedure.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Montgomery Asberg Depression Rating Scale | Trajectories from baseline through 1 month
  depression severity; range 0-60; high score=worse outcome
Quick Inventory of Depressive Symptoms | Trajectories from baseline through 1 month
  Self-reported depression (range: 0-27; higher scores = worse outcome)

SECONDARY OUTCOMES:
Hamilton Depression Rating Scale modified score | Trajectories from baseline through 1 month
  Clinician-rated depression (range: 0-52; higher scores = worse outcome)
Clinical Global Impression Scale--Improvement | Trajectories from baseline through 1 month
  range 1-7 (higher score=worse outcome)
Clinical Global Impression Scale--Severity | Trajectories from baseline through 1 month
  range 1-7 (higher score=worse outcome)
Frequency of scheduled esketamine visits | During first month
  The frequency of scheduled esketamine visits, optimized according to clinicians' judgment of response and patient preferences
Number of patients terminated from esketamine therapy | During first 6 months
  Number with esketamine treatment terminated by the clinic's embedded providers due to lack of clinical response after 1-month of treatment

OTHER OUTCOMES:
Client Satisfaction Questionnaire | Assessment at 'post-CT' timepoint (completed approximately 1 week following randomization)
  self-reported satisfaction with treatment; range 8-32; higher score=better rating
Ease of use | Assessment at 'post-CT' timepoint (completed approximately 1 week following randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Helpfulness | Assessment at 'post-CT' timepoint (completed approximately 1 week following randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Satisfaction with Cognitive Training | Assessment at 'post-CT' timepoint (completed approximately 1 week following randomization)
  self-report slider scale rating; range = 0-100; high score=better rating
Future likelihood of using Cognitive Training | Assessment at 'post-CT' timepoint (completed approximately 1 week following randomization)
  self-report slider scale rating; range = 0-100; high score=better rating

CONTACTS AND LOCATIONS:
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No